CLINICAL TRIAL: NCT01801930
Title: A Phase 1 Study of OCV-C02 in Patients With Advanced or Relapsed Colorectal Cancer Who Are Refractory or Intolerant to Standard Chemotherapy
Brief Title: A Phase 1 Study of OCV-C02 in Patients With Advanced or Relapsed Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 293-12-001; JapicCTI-132075 (Other: Japic)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: OCV-C02; Colorectal Cancer; Antigen specific cancer immunotherapeutic
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose level 1 (Experimental)
  Interventions: Drug: OCV-103 and OCV-104
- Dose level 2 (Experimental)
  Interventions: Drug: OCV-103 and OCV-104
- Dose level 3 (Experimental)
  Interventions: Drug: OCV-103 and OCV-104
- Dose level 4 (Experimental)
  Interventions: Drug: OCV-103 and OCV-104

INTERVENTIONS:
Drug: OCV-103 and OCV-104 — 0.3 mg of each
  Arms: Dose level 1
Drug: OCV-103 and OCV-104 — 1 mg of each
  Arms: Dose level 2
Drug: OCV-103 and OCV-104 — 3 mg of each
  Arms: Dose level 3
Drug: OCV-103 and OCV-104 — 6 mg of each
  Arms: Dose level 4

SUMMARY:
To assess the safety and tolerability of OCV-C02 in Patients With Advanced or Relapsed Colorectal Cancer Who Are Refractory or Intolerant to Standard Chemotherapy

DETAILED DESCRIPTION:
The incidence of dose limiting toxicity (DLT) will be evaluated in cohorts of six patients by starting OCV-C02 administration at dose level 1 (OCV-103 and OCV-104 at 0.3 mg each), increasing the dose to dose level 2 (at 1 mg each), level 3 (at 3 mg each), and then up to dose level 4 (at 6 mg each). Once-weekly administration will be repeated four times in each treatment cycle, and the incidence of DLT from Day 1 to Day 29 will be evaluated.

At the end of Cycle 1, patients who wish to continue OCV-C02 treatment and have provided their written consent will be permitted to continue participation in the trial using the same dosing schedule for each subsequent cycle as that for Cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have human leukocyte antigen (HLA)-A*24:02
* Patients who have histologically-confirmed colorectal cancer (adenocarcinoma)
* Patients with advanced or relapsed colorectal cancer who are refractory or intolerant to standard chemotherapy
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1 at the time of enrollment in the trial.

Exclusion Criteria:

* Patients who are HIV antibody test positive
* Patients with an active infection
* Patients who have or are suspected to have CNS metastasis of colon cancer (such as metastatis of the brain)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (3):
- Japan (3):
  - Nagoya
  - Sunto-gun
  - Tokyo

REFERENCES:
- [Derived] Taniguchi H, Iwasa S, Yamazaki K, Yoshino T, Kiryu C, Naka Y, Liew EL, Sakata Y. Phase 1 study of OCV-C02, a peptide vaccine consisting of two peptide epitopes for refractory metastatic colorectal cancer. Cancer Sci. 2017 May;108(5):1013-1021. doi: 10.1111/cas.13227. Epub 2017 May 11. PMID 28266765

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: OCV-103 and OCV-104 (0.3 mg of each)
  One cycle was defined as 28 days of treatment. Each subject received subcutaneous injections on Days 1, 8, 15, and 22 of each cycle.
- Dose Level 2: OCV-103 and OCV-104 (1 mg of each)
  One cycle was defined as 28 days of treatment. Each subject received subcutaneous injections on Days 1, 8, 15, and 22 of each cycle.
- Dose Level 3: OCV-103 and OCV-104 (3 mg of each)
  One cycle was defined as 28 days of treatment. Each subject received subcutaneous injections on Days 1, 8, 15, and 22 of each cycle.
- Dose Level 4: OCV-103 and OCV-104 (6 mg of each)
  One cycle was defined as 28 days of treatment. Each subject received subcutaneous injections on Days 1, 8, 15, and 22 of each cycle.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6
Not completed — Clear progression of the primary disease is observed | 6 | 5 | 6 | 6
Not completed — DLT occurs | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 3 | 3 | 15
  >=65 years | 2 | 1 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (9.0) | 54.8 (10.2) | 65.8 (9.8) | 63.3 (10.1) | 60.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 3 | 8
  Male | 4 | 5 | 4 | 3 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 6 | 6 | 6 | 6 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: [Definition of DLT]
  Any of the following adverse events (AEs) that occurred by Day 29 of Cycle 1 and for which a causal relationship to OCV-C02 could not be ruled out:
  * Grade 3 or higher non-hematological toxicities (except for injection site reaction and laboratory abnormalities lasting < 7 days without clinical symptoms)
  * The following hematological toxicities: Grade 4 or higher anemia, Grade 4 or higher neutropenia or lymphocytopenia lasting 7 days, Grade 3 or higher febrile neutropenia, Grade 4 or higher platelet count decreased.
  The severity of AEs was graded in accordance with Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Japanese version).
  In addition, a DLT-equivalent treatment-emergent adverse event (TEAE) was defined as a DLT occurred during the extend treatment period (at Cycle 2 and thereafter).
Time Frame: Day 29
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With CTCAE Grade 3 or Higher TEAEs
Description: The severity (grade) of an AE was evaluated using the 5-point scale from Grade 1 to Grade 5 in accordance with CTCAE version 4.0 (Japanese version) , where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE.
Time Frame: From the start of the study drug administration until the completion of the post-treatment observation (28 days after the last administration)
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 3 | 4 | 1 | 3

3. Secondary Outcome: Tumor Response Rate in Cycle 1
Description: Tumor response was graded in accordance with the new Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
  Complete Response (CR): Disappearance of all target lesions (any malignant lymph nodes selected as target lesions must have a reduction in the minor axis to <10 mm) Partial Response (PR): At least a 30% decrease in the diameter sum of the target lesions as compared with the diameter sum at screening Progressive Disease (PD): At least a 20% increase in the diameter sum of the target lesions as compared with the smallest diameter sum recorded after the start of treatment, and at least 5 mm increase in the absolute increase of at least 5 mm Stable Disease (SD): Neither tumor shrinkage equivalent to PR nor tumor enlargement equivalent to PD Not Evaluable (NE): No examination is feasible or the tumor response cannot be considered as any of CR, PR, PD, and SD
Time Frame: Day 29
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants
  CR | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0
  SD | 66.7 | 16.7 | 83.3 | 66.7
  PD | 33.3 | 83.3 | 16.7 | 33.3
  NE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the start of the study drug administration until the completion of the post-treatment observation (28 days after the last administration)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 1/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=6) | Dose Level 3 (N=6) | Dose Level 4 (N=6)
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bile duct stenosi (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=6) | Dose Level 3 (N=6) | Dose Level 4 (N=6)
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 1 | 3 | 1
Malaise (General disorders) | 2 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 0
Induration (General disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 1
Blood urine present (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No